CLINICAL TRIAL: NCT02078726
Title: Role of Glucagon in Outpatient Colonoscopy? A Prospective Double-Blind Randomized Controlled Trial
Brief Title: Glucagon Use in Colonoscopies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 14-13185
Record Dates: First submitted 2014-02-24; First posted 2014-03-05 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Colon Cancer
Keywords: glucagon, screening colonoscopy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucagon (Active Comparator): 1 mg glucagon given during colonoscopy through an IV
  Interventions: Drug: Glucagon
- Placebo (Placebo Comparator): 1 mL normal saline given during colonoscopy through an IV
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon — glucagon (hormone produced by the body) administered through IV

SUMMARY:
The investigators believe that glucagon therapy will have a positive impact on key parameters of colonoscopy such as cecal intubation time, withdrawal time, total procedure time, adenoma detection rate, endoscopist's assessment of the difficulty of the procedure, patient comfort, and patient's willingness to undergo a repeat colonoscopy.

DETAILED DESCRIPTION:
Glucagon transiently decreases peristalsis of smooth muscle in the gastrointestinal tract. It is widely used by radiologists to improve diagnostic yields of upper and lower GI barium contrast examinations. Glucagon is also routinely administered intravenously for all endoscopic retrograde cholangiopancreatography (ERCP) throughout the United States to facilitate canulation of the duodenal papilla and sphincterotomy. Glucagon has been used at the dose of 1-3 mg intravenously by Dr. John Cello in over 5000 ERCP examinations. The role of glucagon in facilitating colonoscopy remains controversial however and is not considered "routine". Several studies have evaluated the effect of glucagon on colonoscopy with varying results. No large scale randomized controlled trial has been performed to conclusively establish the effect of routine glucagon administration prior to colonoscopy. The investigators plan to carry out a randomized double blind, placebo controlled trial that studies key parameters of a colonoscopy such as cecal intubation time, withdrawal time, total procedure time, adenoma detection rate, endoscopist's assessment of the difficulty of the procedure, patient comfort, and patient's willingness to undergo a repeat colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Any subject who has already been already cleared for and scheduled to undergo colonoscopy at SFGH endoscopy center.

Exclusion Criteria:

1. Refusal to give informed consent.
2. Age <18 or >70.
3. Prior intra-abdominal surgery
4. Diabetes
5. Pheochromocytoma
6. Insulinoma
7. Liver disease (Child-Pugh Score >6)
8. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Cello, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Result] Anupam Aditi, Trilokesh Dey Kidambi, Angel Espinoza, Nicholas Crowley, Alex Rodas, John Patrick Cello. Glucagon Shortens Cecal Intubation Time and Total Procedure Time During Colonoscopy: A Prospective, Double-Blind Placebo Controlled Randomized Trial. Biomedical Journal of Scientific & Technical Research. 2019; 22(2).

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucagon: 1 mg glucagon given during colonoscopy
  Glucagon: glucagon (hormone produced by the body)
- Placebo: 1 mL normal saline
  Placebo
Period: Overall Study
Arm/Group | Glucagon | Placebo
Started | 64 | 36
Completed | 64 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glucagon | Placebo | Total
Number analyzed (Participants) | 64 | 36 | 100
Age, Categorical [Count of Participants; unit: Participants] — between 18 and 65
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 64 | 36 | 100
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 19 | 49
  Male | 34 | 17 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 30 | 12 | 42
  Hispanic | 16 | 9 | 25
  Caucasian | 14 | 9 | 23
  African American | 4 | 5 | 9
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 64 | 36 | 100
Diabetes [Count of Participants; unit: Participants] | 18 | 8 | 26
Tobacco use [Count of Participants; unit: Participants] | 21 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Detection Rate (ADR) During Colonoscopy Procedure
Description: ADR was defined as the percentage of participants with at least one traditional adenoma (including tubular or villous adenomas, and adenomas with high grade dysplasia or adenocarcinoma) of any size.
Time Frame: During colonoscopy procedure (an average of 1139 seconds for Glucagon Arm and 1353 seconds for Placebo Arm)
Measure: Number; unit: percentage of participants
Arm/Group | Glucagon | Placebo
Number analyzed (Participants) | 64 | 36
percentage of participants | 43.75 | 33.33

ADVERSE EVENTS:
Time Frame: During colonoscopy procedure (an average of 1139 seconds for Glucagon Arm and 1353 seconds for Placebo Arm)
Arm/Group | Glucagon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/36
Other Adverse Events (participants affected / at risk) | 0/64 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT02078726/Prot_SAP_ICF_001.pdf